CLINICAL TRIAL: NCT02333838
Title: Reduced Toxicity Conditioning Prior to Unrelated Cord Cell Transplantation for High Risk Myeloid Malignancies
Acronym: TBF-Cord
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P130916; 2014-002109-39 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2015-01-07 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Myeloid
Keywords: Cord Cell Transplantation; High risk myeloid malignancies
MeSH Terms: conditions — Leukemia, Myeloid | interventions — Thiotepa; fludarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced toxicity conditioning regimen (Experimental): Reduced toxicity conditioning regimen (thiotepa, busulfan, fludarabine and ATG) followed by unrelated cord blood allogeneic stem cell transplant for high risk myeloïd malignancies.
  The conditioning regimen will include:
  * IV Thiotepa (5 mg/Kg/day for 2 days) (Day -7 and -6)
  * IV fludarabine (40 mg/m²/day for 4 days) (from Day-5 to day -2)
  * IV Busulfan (Busilvex 130 mg/m2/day for 3 days) (Day-5, -4 and -3)
  * IV Anti-thymocyte globuline (Thymogobuline®, 2.5 mg/kg/day for 2 days) (Day-3 and -2)
  In patient with co-morbidities and/or older than 60 years, conditioning could be reduced after consulting the coordinator of the study:
  * IV Thiotepa (5 mg/Kg/day for 2 days) (Day -6)
  * IV fludarabine (40 mg/m²/day for 4 days) (from Day-5 to day -2)
  * IV Busulfan (Busilvex 100 mg/m2/day for 3 days) (Day-5, -4 and -3)
  * IV Anti-thymocyte globuline (Thymogobuline®, 2.5 mg/kg/day for 2 days) (Day-3 and -2)
  Interventions: Drug: IV Thiotepa; Drug: IV Fludarabine; Drug: IV Busulfan; Drug: IV Anti-thymocyte globuline

INTERVENTIONS:
Drug: IV Thiotepa — IV Thiotepa (5 mg/Kg/day for 2 days) (Day -7 and -6) or IV Thiotepa (5 mg/Kg/day for 2 days) (Day -6)
  Other Names: Thiotepa
Drug: IV Fludarabine — IV fludarabine (40 mg/m²/day for 4 days) (from Day-5 to day -2)
  Other Names: Fludarabine
Drug: IV Busulfan — (Busilvex 130 mg/m2/day for 3 days) (Day-5, -4 and -3) or (Busilvex 100 mg/m2/day for 3 days) (Day-5, -4 and -3)
  Other Names: Busulfan
Drug: IV Anti-thymocyte globuline — (Thymogobuline®, 2.5 mg/kg/day for 2 days) (Day-3 and -2)
  Other Names: Anti-thymocyte globuline

SUMMARY:
Allogeneic cord blood stem cell transplantation is a potentially curative therapy for patients with haematological malignancies. We have extensive experience with the use of Cord Blood Transplantation (CBT) in patients with advanced myeloid malignancies. In adults however, the 40% Non-Relapse Mortality (NRM) rate observed after CBT conditioned with a myeloablative conditioning has encouraged the development of CBT with Reduced Intensity Conditioning (RIC). Our previous national CBT protocol (the Minicord French protocol - NCT00797758) showed that RIC CBT can reduce NRM, but relapse remains the main post-transplant event (>30% at one year). Thus, the development of reduced toxicity rather than RIC conditioning for CBT is warranted in order to improve the outcome of such transplants by limiting NRM and reducing relapse rate. The Fludarabine, ATG and intensified doses of IV Busulfan (9.6 mg/Kg total dose) regimen is a well-established preparative regimen for reduced-intensity/toxicity conditioning prior to allogeneic stem cell transplantation using peripheral blood stem cells mobilized with G-CSF (ClinicalTrials.gov Identifier: NCT00841724). However, such regimen is likely not sufficient to allow for CB cell engraftment. Thiotepa is an alkylating and radio-mimetic agent with a large anti-tumor activity including leukemic cells, the ability to cross the blood-brain barrier and to improve engraftment of hematopoietic stem cells. This drug has been combined to usual conditioning regimen without increasing the toxicity but improving the engraftment rate and potentially reducing the relapse rate. Thus, in the context of adult CBT for high risk myeloid malignancies, we propose to prospectively evaluate a reduced toxicity conditioning based on the association of Thiotepa, Fludarabine, IV Busulfan and ATG with the objective to achieve acceptable NRM rates, and to allow for improved anti-leukemic control based on the cytotoxic component of the conditioning regimen itself, while waiting for the long term immune-mediated disease control (GVL effect).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 65 years
* Patients diagnosed with one of the following diseases (validation of the indication of allogeneic

HSCT with an alternative source of hematopoietic stem cells by centers' local RCP):

* Acute myelogenous leukemia (AML) with intermediate or high risk features ((≥ intermediate risk 1) in CR1 or above according to centers' decision
* Myelodysplastic syndromes with International Prognostic Scoring System (IPSS) score ³ 2 (cf. appendix 3) or with symptomatic pancytopenia according to centers' decision
* Chronic myelomonocytic leukemia (CMML)
* Both MDS and CMML should have ≤ 10% blasts at transplantation
* Absence of a matched sibling or unrelated donor (10/10 or 9/10 if mismatch on HLA Cw, based on each center's donor selection criteria)
* Cord blood units must be matched with patient at 4, 5, or 6/6 HLA loci, (class I antigenic & class II allelic level)with a minimum of 3.5 x 10^7 TNC/kg recipient body weight in the pre-thawed fraction and with ≥2.5x10^7 TNC/kg for the richest cord blood unit and ≥ 1.5x10^7 TNC/kg for the poorest blood unit in case of 2 cord blood units
* Performance status : OMS score ≤ 1 (cf. appendix 5)
* Cardiac function - left ventricular ejection fraction ≥ 45%.
* Pulmonary function - diffusion capacity of at least 50% predicted.
* Serum creatinine clearance 0 ml/min.
* SGPT 4x normal , serum bilirubin < 2 x normal.
* Written informed consent.
* Progestative treatment for women with persisting menstrual periods

Exclusion Criteria:

* Presence of a matched sibling or unrelated available donor (10/10 or 9/10 if mismatch on HLA Cw in centers performing 9/10 HLA mismatched transplants)
* Active infection at time of conditioning. In case of uncertainty regarding whether a previous infection is resolved or not, this will be discussed with the PI on a case by case basis.
* Pregnancy in women with child bearing potential (pregnancy test performed within 2-4 weeks of study entry).
* HIV positive
* Active CNS leukemia
* Chronic or active Hepatitis B or Hepatitis C. If questions about liver health discuss with PI and strongly consider liver biopsy.
* Poor performance status : OMS score > 1
* Life expectancy is severely limited by concomitant illness and expected to be <12 weeks.
* Left ventricular ejection fraction <45%. Uncontrolled arrhythmias or symptomatic cardiac disease.
* Symptomatic pulmonary disease. FEV1, FVC and DLCO <50% of expected corrected for hemoglobin.
* Serum creatinine clearance (Crockoft) below 50 mL/m per 1.73 m² or requiring dialysis
* Vaccination with alive vaccine (virus or bacteria) < 3 months
* Fludarabine contra-indication
* Thymoglobuline contra-indication
* Patient under guardianship or curatorship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of NRM at 12 months after transplantation | 12 months after transplantation
  Cumulative incidence of NRM at 12 months after transplantation : Safety and efficacy of the pre-transplant reduced toxicity conditioning regimen

SECONDARY OUTCOMES:
Incidence of engraftment after transplantation | 12 months after transplantation
  Incidence of neutrophil engraftment (day and proportion of patients reaching neutrophils >0.5x109/L); and platelets recovery (day and proportion of patients reaching platelets > 20 x 109 / L without transfusion) after transplantation
Incidence and severity of acute GVHD | 6 months after transplantation
  Incidence and severity of acute GVHD (diagnosed and graded as standard criteria)
Incidence and severity of chronic GVHD | 12 months after transplantation
  Incidence and severity of chronic GVHD (diagnosed and graded as standard criteria detailed )
Rate of disease relapse at one year after transplantation | 12 months after transplantation
  Incidence of disease relapse at one year after transplantation (relapse is defined on the basis of morphologica evidence of leukemic cells in the bone marrow or other sites)
Quality of life | 12 months after transplantation
  Evaluation of the quality of life (using a french translation of the FACT-BMT (version 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Thérèse RUBIO, Principal Investigator — CHRU Nancy
Locations (1):
- Hôpital de Brabois, Hématologie Clinique et thérapie cellulaire, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Rocha V, Labopin M, Sanz G, Arcese W, Schwerdtfeger R, Bosi A, Jacobsen N, Ruutu T, de Lima M, Finke J, Frassoni F, Gluckman E; Acute Leukemia Working Party of European Blood and Marrow Transplant Group; Eurocord-Netcord Registry. Transplants of umbilical-cord blood or bone marrow from unrelated donors in adults with acute leukemia. N Engl J Med. 2004 Nov 25;351(22):2276-85. doi: 10.1056/NEJMoa041469. PMID 15564544
- [Background] Arcese W, Rocha V, Labopin M, Sanz G, Iori AP, de Lima M, Sirvent A, Busca A, Asano S, Ionescu I, Wernet P, Gluckman E; Eurocord-Netcord Transplant group. Unrelated cord blood transplants in adults with hematologic malignancies. Haematologica. 2006 Feb;91(2):223-30. PMID 16461307
- [Background] Atsuta Y, Suzuki R, Nagamura-Inoue T, Taniguchi S, Takahashi S, Kai S, Sakamaki H, Kouzai Y, Kasai M, Fukuda T, Azuma H, Takanashi M, Okamoto S, Tsuchida M, Kawa K, Morishima Y, Kodera Y, Kato S; Japan Cord Blood Bank Network. Disease-specific analyses of unrelated cord blood transplantation compared with unrelated bone marrow transplantation in adult patients with acute leukemia. Blood. 2009 Feb 19;113(8):1631-8. doi: 10.1182/blood-2008-03-147041. Epub 2008 Dec 22. PMID 19104080
- [Background] Eapen M, Rocha V, Sanz G, Scaradavou A, Zhang MJ, Arcese W, Sirvent A, Champlin RE, Chao N, Gee AP, Isola L, Laughlin MJ, Marks DI, Nabhan S, Ruggeri A, Soiffer R, Horowitz MM, Gluckman E, Wagner JE; Center for International Blood and Marrow Transplant Research; Acute Leukemia Working Party Eurocord (the European Group for Blood Marrow Transplantation); National Cord Blood Program of the New York Blood Center. Effect of graft source on unrelated donor haemopoietic stem-cell transplantation in adults with acute leukaemia: a retrospective analysis. Lancet Oncol. 2010 Jul;11(7):653-60. doi: 10.1016/S1470-2045(10)70127-3. PMID 20558104